CLINICAL TRIAL: NCT05193097
Title: Vasopressor Preload Modulation During General Anaesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jakob Højlund (Other)
Responsible Party: Sponsor-Investigator, Jakob Højlund, Assistant professor, consultant, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: H-21032981
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia
Keywords: monitoring; cardiac output; perfusion index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Is is debated whether administration of pure vasopressor may augment cardiac output (CO) by means of preload modulation. We wish to test this in 20 patients under general anesthesia, with preload dependency induced by head-up-tilt and preload modulation with infusion of phenylephrine. To document any changes in CO the patients will be monitored by Lithium dilution method. Furthermore we will monitor changes in peripheral perfusion index and test the ability of this non-invasive modality to track changes in CO.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery under general anesthesia

Exclusion Criteria:

* atrial fibrillation
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patient with planned surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiac output | 30 minutes
Changes in peripheral perfusion index | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Højlund, MD, Principal Investigator — Hvidovre University Hospital

REFERENCES:
- [Derived] Hojlund J, Cihoric M, Foss NB. Vasoconstriction with phenylephrine increases cardiac output in preload dependent patients. J Clin Monit Comput. 2024 Oct;38(5):997-1002. doi: 10.1007/s10877-024-01186-7. Epub 2024 Jun 21. PMID 38907106